CLINICAL TRIAL: NCT02013141
Title: An Open-Label Study of the Pharmacokinetics of a Single Dose of Telavancin in Pediatric Subjects Aged 12 Months to 17 Years
Brief Title: Telavancin Pediatric PK Study (Ages >12 Months to 17 Years)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: FDA waived the pediatric study requirement for this application
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0101
Record Dates: First submitted 2013-12-11; First posted 2013-12-17 (Estimated); Results first posted 2024-06-24 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-01

CONDITIONS: Gram-Positive Bacterial Infections
Keywords: Gram positive bacteria; Telavancin; VIBATIV; Pediatric; Pharmacokinetics
MeSH Terms: conditions — Gram-Positive Bacterial Infections | interventions — telavancin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Telavancin (Experimental): Telavancin 10 mg/kg IV administered over approximately 60 minutes one time.
  Interventions: Drug: Telavancin

INTERVENTIONS:
Drug: Telavancin
  Other Names: VIBATIV; TD-6424

SUMMARY:
This is a multicenter, open-label, single-dose pharmacokinetic (PK) study. Infants, children, and adolescents will receive a single 10 mg/kg dose of telavancin infused intravenously (IV) over 60 minutes

DETAILED DESCRIPTION:
This is a multicenter, open-label, single-dose pharmacokinetic (PK) study. Infants, children, and adolescents will receive a single 10 mg/kg dose of telavancin infused intravenously (IV) over 60 minutes in male or female infants, children, and adolescents (> 12 months to 17 years, inclusive) who require systemic antibiotic therapy for the treatment or prevention of a known or suspected bacterial infection.

Blood samples for PK assessment will be taken as follows: 1.0 hour (±5 min), 1.5 hours (±5 min), 2 hours (±5 min), 6 hours (±30 min), 12 hours (±30 min) and 24 hours (±30 minutes) after the beginning of the infusion. The timing of PK sampling may be optimized after the completion of the older age groups (Cohorts 1-3) to assure that the minimum numbers of samples are collected in the youngest age group > 12months to < 24 months. Plasma exposures that will be compared to adult exposures are the primary assessment for this study.

Subject safety will be monitored during the study using standard measures, including physical examinations, vital signs, 12-lead ECGs, clinical laboratory assessments, urinalysis, concomitant medication usage, and adverse event reporting.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 12 months to 17 years of age (inclusive)
2. Subject's weight is within the 3rd to 97th percentile (inclusive) for age and sex.
3. Written informed consent and assent (if appropriate for older age groups) has been obtained per institutional review board (IRB) policy and requirements, consistent with ICH guidelines.
4. Male and female subjects of reproductive potential (i.e., post-pubertal males and post-menarche females) must agree to use a highly effective method of contraception throughout study period and for 30 days after administration of study drug. A highly effective method of birth control is defined as one that results in a low failure rate (i.e., <1% per year) when used consistently and correctly, such as condom + diaphragm, condom + spermicide, diaphragm + spermicide; or intrauterine device (IUD) with documented failure rate of <1% per year; or oral/injectable/implanted hormonal contraceptives used in combination with an additional double-barrier method; or sexual abstinence.
5. Female subjects who are post menarche are required to have a negative serum pregnancy test before the administration of study drug.
6. Subject requires or recently completed systemic antibiotic therapy for the treatment or prevention of a known or suspected bacterial infection. If completed, the last administered dose of systemic antibiotic must be within 24 hours of enrollment.

Exclusion Criteria:

1. Subject has an estimated creatinine clearance <50 mL/min/1.73 m2 (Schwartz equation).
2. Any clinically significant abnormal laboratory value, including hematology, chemistry, or urinalysis that in the judgement of the investigator would make it difficult to assess the pharmacokinetic profile and safety of a single dose of telavancin or would compromise the safety of the subject.
3. Any clinically significant medical history, abnormal physical examination finding, or vital sign measurement, including evidence of hemodynamic instability or significant collections of fluid outside normal vascular and tissue compartments (e.g., large pleural effusions, ascites), that in the judgement of the investigator would make it difficult to assess the pharmacokinetic profile or safety of a single dose of telavancin or would compromise the safety of the subject.
4. Subject has clinically relevant cardiac abnormality, in the opinion of the investigator, such as:

   1. A mean QTcF >440 msec, congenital long QT syndrome, second or third degree heart block at rest.
   2. Hemodynamically significant heart disease, eg, hemodynamically unstable congenital heart defect, uncompensated heart failure, uncorrected abnormal calcium, hyperkalemia, or any other unstable cardiac condition.
   3. An arrhythmic heart condition requiring medical therapy
5. Subject is receiving an anticoagulant AND requires specific coagulation testing (Prothrombin Time/International Normalized Ratio, Activated Partial Thromboplastin Time, Activated Clotting Time, or Coagulation Based Factor X Activity Assay) within 24 hours of receiving the telavancin dose. NOTE: Although telavancin does not interfere with coagulation, it interferes with some assays used to monitor coagulation.
6. Subjects who are receiving concomitant vancomycin treatment should not be assessed for vancomycin serum concentrations within 24 hours of receiving the Telavancin dose. NOTE: Telavancin might interfere with some Vancomycin therapeutic drug monitoring assays. Caution should be exercised when interpreting vancomycin drug monitoring levels in the presence of telavancin.
7. Subject has a history of allergies or hypersensitivities to glycopeptide antibiotics (e.g., vancomycin), telavancin, or the formulation excipients.
8. Subject requires, or is anticipated to require, concomitant [within 24 hours before or 24 hours following the single dose of study medication (telavancin)] administration of agents that in the clinical judgment of the investigator increase the risk of torsade de pointes.
9. Subject is considered unlikely to comply with the study procedures.
10. Subject was treated with an investigational drug within 30 days or five half-lives, whichever is longer, before study entry.
11. Subject has any other condition that, in the opinion of an investigator, would confound or interfere with evaluation of safety of the investigational drug, or prevent compliance with the study protocol.

Ages: 12 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital San Diego, San Diego, California
  - Children's Mercy Hospital, Kansas City, Missouri
  - Rutgers-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Toledo Children's Hospital, Toledo, Ohio

REFERENCES:
- [Derived] Bradley JS, Goldman JL, James LP, Kaelin B, Gibson BHY, Arrieta A. Pharmacokinetics and safety of a single dose of telavancin in pediatric subjects 2-17 years of age. Antimicrob Agents Chemother. 2023 Nov 15;67(11):e0098723. doi: 10.1128/aac.00987-23. Epub 2023 Oct 10. PMID 37815398

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (Age 12 to 17 Years): Participants 12 to 17 years of age who received 10 mg/kg IV telavancin administered over one hour one time.
- Cohort 2 (Age 6 to 11 Years): Participants 6 to 11 years of age who received 10 mg/kg IV telavancin administered over one hour one time.
- Cohort 3 (Age 2 to 5 Years): Participants 2 to 5 years of age who received 10 mg/kg IV telavancin administered over one hour one time.
Period: Overall Study
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort 2 (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
Started | 14 | 7 | 1
Completed | 14 | 7 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort 2 (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years) | Total
Number analyzed (Participants) | 14 | 7 | 1 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 15.1 (1.69) | 8.57 (2.44) | 2 (NA) — Standard deviation cannot be calculated for a single subject | 12.4 (4.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 1 | 10
  Male | 6 | 6 | 0 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 4 | 4 | 1 | 9
  Ethnicity: Not Hispanic or Latino | 9 | 3 | 0 | 12
  Ethnicity: Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 13 | 7 | 1 | 21
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 64.2 (15.3) | 35.6 (10.5) | 12.3 (NA) — Standard deviation cannot be calculated for a single subject | 52.9 (21.4)
Height [Mean (Standard Deviation); unit: cm] | 165 (11.9) | 136 (13.6) | 81.0 (NA) — Standard deviation cannot be calculated for a single subject | 152 (24.8)
BMI [Mean (Standard Deviation); unit: kg/m2] — Body mass index
  kg/m2 | 23.2 (3.63) | 18.8 (2.11) | 18.7 (NA) — Standard deviation cannot be calculated for a single subject | 21.6 (3.86)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics- Area Under the Curve Extrapolated to Infinity for the Plasma Concentration Versus Time Curves for Telavancin
Description: Plasma telavancin concentrations were measured at 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours following IV infusion of telavancin, and area under the curve extrapolated to infinity was calculated for the plasma concentration versus time curves for telavancin following a single 10 mg/kg IV dose.
Time Frame: 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours
Population: Pharmacokinetic population- one subject from Cohort 1 and one subject from Cohort 2 were excluded due to lack of pharmacokinetic plasma samples at >1 time point
Measure: Mean (Standard Deviation); unit: h*mcg/ml
Groups:
- Cohort (Age 6 to 11 Years): Participants 6 to 11 years of age who received 10 mg/kg IV telavancin administered over one hour one time.
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
Number analyzed (Participants) | 13 | 6 | 1
h*mcg/ml | 345 (58.8) | 351 (79.7) | 229 (NA) — Standard deviation cannot be calculated for a single subject

2. Primary Outcome: Pharmacokinetics- Maximum Plasma Concentration of Telavancin
Description: Plasma telavancin concentrations were measured at 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours following IV infusion of telavancin to provide the maximum plasma concentration of telavancin following a single 10 mg/kg IV dose.
Time Frame: 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
Number analyzed (Participants) | 13 | 6 | 1
mcg/mL | 58.3 (8.40) | 60.1 (11.9) | 53.1 (NA) — Standard deviation cannot be calculated for a single subject

3. Primary Outcome: Pharmacokinetics- Time to Maximum Plasma Telavancin Concentration
Description: Plasma telavancin concentrations were measured at 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours following IV infusion of telavancin to provide the time to maximum plasma concentration of telavancin following a single 10 mg/kg IV dose.
Time Frame: 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
Number analyzed (Participants) | 13 | 6 | 1
hours | 1.02 [1.00 to 1.55] | 1.09 [1.00 to 1.32] | 1.18 [1.18 to 1.18]

4. Primary Outcome: Pharmacokinetics- Terminal Elimination Half-life for Plasma Telavancin
Description: Plasma telavancin concentrations were measured at 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours following IV infusion of telavancin, and the terminal elimination half-life was calculated from the plasma concentration versus time curves for telavancin following a single 10 mg/kg IV dose.
Time Frame: 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
Number analyzed (Participants) | 13 | 6 | 1
hours | 5.60 (1.01) | 5.19 (0.751) | 2.73 (NA) — Standard deviation cannot be calculated for a single subject

5. Primary Outcome: Pharmacokinetics- Area Under the Curve From Time Zero to the Last Sample for the Telavancin Plasma Concentration Versus Time Curve
Description: Plasma telavancin concentrations were measured at 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours following IV infusion of telavancin, and area under the curve from time zero to the last sample was calculated for the plasma concentration versus time curves for telavancin following a single 10 mg/kg IV dose.
Time Frame: 1.0, 1.5, 2.0, 6.0, 12.0, 24.0 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*mcg/mL
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
Number analyzed (Participants) | 13 | 6 | 1
h*mcg/mL | 326 (50.0) | 333 (74.2) | 228 (NA) — Standard deviation cannot be calculated for a single subject

6. Secondary Outcome: Safety- Number of Treatment-emergent Adverse Events.
Description: Treatment-emergent adverse events were monitored during the study using standard measures, including physical examinations, vital signs, 12-lead ECGs, clinical laboratory assessments, urinalysis, and symptom reporting.
Time Frame: Day 0 (screening) through follow-up on Day 8 (+/- 1 day)
Population: Safety population- includes all 22 study participants
Measure: Number; unit: events
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
Number analyzed (Participants) | 14 | 7 | 1
events | 16 | 11 | 0

7. Secondary Outcome: Safety- Number of Subjects With Treatment-emergent Adverse Events
Description: as for outcome 6
Time Frame: Day 0 (screening) through follow-up on Day 8 (+/- 1 day)
Population: Safety population- includes all 22 study participants
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
Number analyzed (Participants) | 14 | 7 | 1
Participants | 6 | 4 | 0

ADVERSE EVENTS:
Time Frame: Eight days following telavancin administration
Description: Treatment-emergent adverse events were monitored during the study using standard measures, including physical examinations, vital signs, 12-lead ECGs, clinical laboratory assessments, urinalysis, and symptom reporting.
Arm/Group | Cohort 1 (Age 12 to 17 Years) | Cohort (Age 6 to 11 Years) | Cohort 3 (Age 2 to 5 Years)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/7 | 0/1
Other Adverse Events (participants affected / at risk) | 6/14 | 4/7 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (Age 12 to 17 Years) (N=14) | Cohort (Age 6 to 11 Years) (N=7) | Cohort 3 (Age 2 to 5 Years) (N=1)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (3) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Information on the pharmacokinetics and safety of a single dose of telavancin in subjects aged 2 to 5 years is limited as Cohort 3 only enrolled 1 participant due to early termination of the study. No infants were enrolled due to early termination of the study, and therefore, no information is available on the pharmacokinetics and safety of a single dose of telavancin in infants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period up to 90 days. The sponsor can require changes to the communication but cannot extend the embargo beyond the 90 days.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-26): https://cdn.clinicaltrials.gov/large-docs/41/NCT02013141/Prot_SAP_000.pdf